CLINICAL TRIAL: NCT02772289
Title: A Phase II, Randomized, Double-Blind, Placebo-Controlled Study of the Efficacy and Safety of Perinatal Tissue Mesenchyme Stem Cells in the Treatment for Caesarean Section Scars
Brief Title: Perinatal Tissue Mesenchyme Stem Cells in the Treatment for Caesarean Section Scars
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Maternal and Child Health Hospital of Foshan (Other)
Responsible Party: Principal Investigator, Zhengping Liu, MD, Director, Maternal and Child Health Hospital of Foshan
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MCHHFoshan-1602
Record Dates: First submitted 2016-05-10; First posted 2016-05-13 (Estimated); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Cicatrix
Keywords: Mesenchyme Stem Cells; Cesarean Section; Scars
MeSH Terms: conditions — Cicatrix | interventions — Population Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Mesenchymal Stem Cells low-dose group (Experimental): Target dose of 3 million Mesenchymal Stem Cells
  Interventions: Biological: Mesenchyme Stem Cells low-dose group
- Mesenchymal Stem Cells high-dose group (Experimental): Target dose of 6 million Mesenchymal Stem Cells
  Interventions: Biological: Mesenchyme Stem Cells high-dose group
- Placebo (Placebo Comparator): Placebo without Mesenchyme Stem Cells
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Mesenchyme Stem Cells low-dose group — Participants will receive transdermal one dose of 1*10^6 cells of Perinatal Tissue Mesenchyme Stem Cells in the gel once a day for continuous three days and then receive transdermal placebo without of Perinatal Tissue Mesenchyme Stem Cells in the gel once a day for continuous next three days.
  Arms: Mesenchymal Stem Cells low-dose group
Biological: Mesenchyme Stem Cells high-dose group — Participants will receive transdermal one dose of 1*10^6 cells of Perinatal Tissue Mesenchyme Stem Cells in the gel once a day for continuous six days.
  Arms: Mesenchymal Stem Cells high-dose group
Biological: Placebo — Participants will receive transdermal placebo without of Perinatal Tissue Mesenchyme Stem Cells in the gel once a day for continuous six days.
  Arms: Placebo

SUMMARY:
The study is to investigate the efficacy and safety of perinatal tissue mesenchyme stem cells treatment on the appearance of a caesarean scar as compared to a similar untreated scar.

DETAILED DESCRIPTION:
Nowadays, cesarean is one of the most common surgical interventions and its prevalence has increased in most countries in the recent years. Delay in healing of cesarean wound and formation of visible scar are common symptoms of maternal morbidity after cesarean section. These complications affect mother's quality of life due to stress, anxiety, delay in mother's ability and health recovery, and also they are associated with additional cost as a result of the increased need for wide spectrum antibiotics and sometimes hospitalization and repeated repair of wound. Improve the final aspect of would and visible scars, have been a challenge for medicine. Mesenchymal stem cells (MSC) are a population of pluripotent stem cells that are self-renewing and capable of differentiating into canonical cells of the mesenchyme. Recently, stem cells have been applied to regenerative medicine, even for internal organs such as blood vessels, nerves, and heart.

The study is to investigate the efficacy and safety of perinatal tissue mesenchyme stem cells treatment on the appearance of a caesarean scar as compared to a similar untreated scar. This is a randomized, double-blind, placebo-controlled clinical trial designed to investigate the efficacy and safety of perinatal tissue mesenchyme stem cells (MSC) treatment on the appearance of a caesarean scar as compared to a similar untreated scar. A total of ninety (90) participants will be randomized (1:1:1) to receive MSC or placebo. All of participants will be undergoing delivery by lower segment caesarean section through a transverse abdominal incision, and there will be no clear indication for a particular surgical technique or material to be used. In low-dose MSC group, participants will receive transdermal one dose of 1*10^6 cells of Perinatal Tissue Mesenchyme Stem Cells in the gel once a day for continuous three days and then receive transdermal placebo without of Perinatal Tissue Mesenchyme Stem Cells in the gel once a day for continuous next three days; In high-dose MSC group, participants will receive transdermal one dose of 1*10^6 cells of Perinatal Tissue Mesenchyme Stem Cells in the gel once a day for continuous six days; And in placebo group, participants will receive transdermal placebo without of Perinatal Tissue Mesenchyme Stem Cells in the gel once a day for continuous six days. After randomization, baseline data, and transdermal treatment, participants will be followed up at 1 month, 3 months and 6 months. For the purpose of the endpoint analysis and safety evaluations, the investigators will utilize an "intention-to-treat" study population.

ELIGIBILITY:
Inclusion Criteria:

* Primiparous women receiving cesarean delivery
* Ages between 21-35 years
* Gestation ages ≥ 37 weeks and < 42 weeks
* Willing to give and sign an informed consent form and a photographic release form
* Willing to comply with study dosing and complete the entire course of the study

Exclusion Criteria:

* Any systemic uncontrolled disease
* Recent or current cancer
* History or presenting with a keloid formation
* Wounds or local disease in treatment area
* Planning any other cosmetic procedure to the study area during the study period
* Smoking

Ages: 21 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Change of Vancouver Scar Scale (VSS) | 1st, 3rd, 6th month post treatment
  The investigators measured quartile grading scale at 1st, 3rd and 6th months of study and evaluated the change of the scale

SECONDARY OUTCOMES:
Wound healing status | 14 days post surgery
  Wound healing status was assessed using REEDA scale which is based on the amount of redness, edema, ecchymosis, discharge and the approximation of wound edges (each one scored between 0-3); the final score was the sum of the items scores. Lower score indicated better healing.
Erythema measured by reflectance | 1st, 3rd, 6th month post treatment
  measured by reflectance
Pigmentation measured by reflectance | 1st, 3rd, 6th months post treatment
  measured by reflectance
Scar Thickness and Uniformity | 1st, 3rd, 6th month post treatment
  A High Definition Ultrasound (US) device will be used to generate a high resolution image of the skin layers of the treated and non-treated scar in order to measure and compare changes in scar thickness and uniformity.
Change of scar area | 1st, 3rd, 6th month post treatment
  A High Definition Ultrasound (US) device will be used to generate a high resolution image of the skin layers of the treated and non-treated scar in order to measure and compare changes in scar area.
Immunoglobulin concentrations in breast milk | 1st, 3rd, 6th month post treatment
  Breast milk immunoglobulin (IgG, IgA, IgM) and the complement (C3, C4) were detected by transmission immune turbidity method using automatic biochemical analyzer.
Subject's satisfaction | 6th month post treatment
  Subject's satisfaction of the treatment using a Satisfaction Scale as follows: None; Slight; Moderate; Good; Very Good.
Adverse events occurrence | 6 months
  Adverse events will be evaluated since the baseline visit until 6 months after the end of the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Zhengping Liu, MD, Principal Investigator — Maternal and Child Health Hospital of Foshan
Locations (1):
- Maternal and Child Health Hospital of Foshan, Foshan, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Fan D, Zeng M, Xia Q, Wu S, Ye S, Rao J, Lin D, Zhang H, Ma H, Han Z, Guo X, Liu Z. Efficacy and safety of umbilical cord mesenchymal stem cells in treatment of cesarean section skin scars: a randomized clinical trial. Stem Cell Res Ther. 2020 Jun 25;11(1):244. doi: 10.1186/s13287-020-01695-7. PMID 32586366
- [Derived] Fan D, Xia Q, Wu S, Ye S, Liu L, Wang W, Guo X, Liu Z. Mesenchymal stem cells in the treatment of Cesarean section skin scars: study protocol for a randomized, controlled trial. Trials. 2018 Mar 2;19(1):155. doi: 10.1186/s13063-018-2478-x. PMID 29499740